CLINICAL TRIAL: NCT02354963
Title: Follicle Activation in Patients With Poor Ovarian Response Through Fragmentation of the Ovarian Tissue.
Brief Title: Follicular Activation in Poor Responders
Acronym: FAPPOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: César Díaz García (Other)
Responsible Party: Sponsor-Investigator, César Díaz García, PhD, MD, Instituto de Investigacion Sanitaria La Fe
Organization: Instituto de Investigacion Sanitaria La Fe (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAPPOR (2014/0004)
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Infertility
Keywords: Poor ovarian response; Salvador/Warts/Hippo pathway; Follicular activation; Poor ovarian reserve
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (No Intervention): No intervention is performed. Assessment of antral follicle count. IVF treatment.
- Experimental arm (Experimental): Perform intervention described: Laparoscopy. In vitro fragmentation of the ovarian tissue.
  Assessment of antral follicle count. IVF treatment.
  Interventions: Procedure: In vitro fragmentation of the ovarian tissue

INTERVENTIONS:
Procedure: In vitro fragmentation of the ovarian tissue — Unilateral ovarian cortex extraction, in vitro fragmentation and reimplantation.
  Arms: Experimental arm

SUMMARY:
This study aims to assess whether activation of primordial follicles through ovarian cortex fragmentation may increase the number of antral follicles present in the ovary of patients with diminished ovarian reserve. Secondary outcomes include number of oocytes retrieved and pregnancy rates after IVF.

Hypothesis; Evaluate whether the proposed intervention increases the pool of antral follicles (potentially stimulable ones).

DETAILED DESCRIPTION:
Controlled, randomized, assessor-blind clinical trial.

Thirty-six patients of La Fe University Hospital (Valencia), previously confirmed as poor responders according to the European Society of Human Reproduction and Embryology (ESHRE) criteria, will be randomized to two treatment arms:

* Arm 1 (control): no intervention.
* Arm 2 (intervention): ovarian cortex extraction by unilateral laparoscopic biopsy and ovarian tissue fragmentation in aliquots of 1 mm2. These fragments will be grafted under the ovarian cortex and meso-ovarium ipsilateraly.

Subsequently the number of antral follicles in both intervention groups will be compared and also will be the number of antral follicles in the native ovary and the grafted one in each of the patients.

Patients will receive a standard IVF treatment for poor responders according to the protocols of the assisted reproduction unit of La Fe University Hospital.

The final aim is to assess the pregnancy rate in both groups, as well as parameters related to the reproduction technique when required.

ELIGIBILITY:
Inclusion Criteria (must meet one):

* At least two episodes of poor ovarian response (≤ 3 oocytes retrieved with a standard protocol).
* A previous IVF cycle with ≤ 3 oocytes (following a standard stimulation protocol) and presence of an abnormal ovarian reserve test (antral follicle count of ≤ 5 or antimüllerian hormone ≤ 5pm).

Exclusion Criteria (must not meet any):

* Patients under 18 or over 40 years.
* Clinical signs of endometriosis.
* Previous ovarian surgery.
* Genital tract malformations.
* Anovulatory patient (defined by the presence of irregular cycles and serum progesterone ≤ 10 ng / mL on cycle day 21).
* Partner with severe male factor: severe oligoasthenozoospermia, oligoasthenoteratozoospermia and azoospermia.
* All those patients who do not voluntarily give their express written consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-11; Primary Completion 2019-02 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Diaz-Garcia, MD, Principal Investigator — La Fe University Hospital. University of Valencia
Locations (1):
- La Fe University Hospital, Valencia, Spain

REFERENCES:
- [Derived] Diaz-Garcia C, Herraiz S, Pamplona L, Subira J, Soriano MJ, Simon C, Seli E, Pellicer A. Follicular activation in women previously diagnosed with poor ovarian response: a randomized, controlled trial. Fertil Steril. 2022 Apr;117(4):747-755. doi: 10.1016/j.fertnstert.2021.12.034. PMID 35367015

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Perform intervention described: Laparoscopy. In vitro fragmentation of the ovarian tissue.
  Assessment of antral follicle count. IVF treatment.
  In vitro fragmentation of the ovarian tissue: Unilateral ovarian cortex extraction, in vitro fragmentation and reimplantation.
Period: Overall Study
Arm/Group | Control Arm | Experimental Arm
Started | 18 | 16
Completed | 16 | 15
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Two participants in the control group and one in the surgery group were lost after assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Experimental Arm | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36.5 [35 to 38] | 36.5 [34 to 37.7] | 36.5 [36.5 to 36.5]
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Partner's age (years old)
  years | 37 [33 to 42] | 37.5 [37 to 39.7] | 37.3 [37 to 37.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] — Body Mass Index (BMI) was calculated for all the recruited patients according to the formula kg/m^2.
  kg/m^2 | 21 [19.8 to 23.6] | 22.4 [20.2 to 24.0] | 21.7 [21 to 22.4]
Previous gestations [Count of Participants; unit: Participants] | 7 | 6 | 13
Previous deliveries [Count of Participants; unit: Participants] | 1 | 1 | 2
Previous miscarriages [Count of Participants; unit: Participants] | 6 | 5 | 11
Infertility etiology [Count of Participants; unit: Participants]
  Only POR | 16 | 15 | 31
  Tubal factor | 1 | 1 | 2
  Male factor | 1 | 0 | 1
Infertile duration [Mean (Inter-Quartile Range); unit: months] | 36 [36 to 72] | 48 [36 to 87] | 42 [36 to 48]
Baseline Antral Follicle Count (AFC) [Median (Inter-Quartile Range); unit: number of follicles] | 5 [2 to 5] | 4 [2 to 4] | 4.5 [4 to 5]
Baseline AMH [Mean (Inter-Quartile Range); unit: ng/mL] | 0.36 [0.08 to 0.56] | 0.44 [0.18 to 0.50] | 0.4 [0.36 to 0.44]
Number of previous IVF cycles [Count of Participants; unit: Participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Metaphase II (MII)
Description: Number of mature MII oocytes retrieved in the IVF cycles after triggering.
Time Frame: 36 hours after triggering
Population: Of the 18 patients in the initial control group, 2 dropped out of the study (one because she did not want to follow up and the other because she divorced). Of the 16 patients in the experimental group, one patient left the study before treatment because she moved to another city.
Measure: Median (Inter-Quartile Range); unit: Oocytes
Units Other Than Participants: Number of IVF cycles
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of IVF cycles) | 16 | 15
Oocytes | 4 [1 to 8] | 2 [1 to 3]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.302, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Total Antral Follicle Count (AFC) - Initial Measure
Description: AFC assessment was done on day 2-5 of the menstrual cycle. Ultrasound scan was performed using a GE iVoluson (General Electric, Spain) equipped with a 3D vaginal probe (6.5-9MHz). A bilateral two-dimensional scan was performed and the mean of the two largest diameters of each intra-ovarian avascular anechoic image was recorded. Antral follicles with a mean diameter from 2 to 10 mm were counted to establish AFC. Initial data refers to the measure taken before treatment.
Time Frame: Baseline, day 2-5 of the menstrual cycle prior to treatment
Population: Of the 18 patients in the initial control group, 2 dropped out of the study (one because she did not want to follow up and the other because she divorced her husband). Of the 16 patients in the experimental group, one patient left the study before treatment because she moved to another city.
Measure: Median (Inter-Quartile Range); unit: Follicles
Units Other Than Participants: Number of IVF cycles
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of IVF cycles) | 16 | 15
Follicles | 5 [2 to 5] | 4 [2 to 4]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.449, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Total Antral Follicle Count (AFC) - Final
Description: AFC assessment was done on day 2-5 of the menstrual cycle and was followed for 6-month. To determine AFC, ultrasound scan was performed using a GE iVoluson (General Electric, Spain) equipped with a 3D vaginal probe (6.5-9MHz). A bilateral two-dimensional scan was performed and the mean of the two largest diameters of each intra-ovarian avascular anechoic image was recorded. Antral follicles with a mean diameter from 2 to 10 mm were counted to establish AFC. Final measure refers to the AFC count after ovarian fragmentation treatment.
Time Frame: Day 2-5 of the menstrual cycle 6 months after treatment
Population: as for outcome 2
Measure: Mean (Inter-Quartile Range); unit: Follicles
Units Other Than Participants: Number of IVF cycles
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of IVF cycles) | 16 | 15
Follicles | 5 [3 to 6] | 5 [3 to 7]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.021, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Initial Antimüllerian Hormone (AMH) Levels
Description: AMH levels were determined on day 2-5 of the menstrual cycle to establish the initial baseline levels for each patient. A microparticle immunoassay kit integrated in the ABBOTT AxSYM® Plus system and software 5.20 (Abbott Laboratories, Abbot Park, IL, USA) was used to determine AMH levels prior treatment.
Time Frame: Baseline, day 2-5 of the menstrual cycle prior to treatment
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Units Other Than Participants: Number of IVF cycles
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of IVF cycles) | 16 | 15
ng/mL | 0.36 [0.08 to 0.56] | 0.44 [0.18 to 0.50]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.427, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Final AMH Levels
Description: AMH levels were determined using a microparticle immunoassay kit integrated in the ABBOTT AxSYM® Plus system and software 5.20 (Abbott Laboratories, Abbot Park, IL, USA) 6 months after recruitment or basaline assessment.
Time Frame: Day 2-5 of the menstrual cycle 6 months after the treatment
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Units Other Than Participants: Number of IVF cycles
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of IVF cycles) | 16 | 15
ng/mL | 0.35 [0.11 to 0.66] | 0.29 [0.20 to 0.69]
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.496, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Cancelled IVF Cycles
Description: Number of cancelled IVF cycles for low or no response to controlled ovarian stimulation. Cycles were cancelled because of a lack of an adequate follicular formation (one follicle of at least 17 mm) the day of triggering.
Time Frame: End of stimulation cycle (less than or equal to 30 days)
Population: as for outcome 2
Measure: Number; unit: Number of cycles
Units Other Than Participants: Number of IVF cycles
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of IVF cycles) | 16 | 15
Number of cycles | 3 | 2
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.684, Chi-squared; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.13 to 3.68]

7. Secondary Outcome: Fertilization Rate
Description: All the mature oocytes retrieved were inseminated by intracytoplasmic sperm injection (ICSI). Percentage of successfully fertilized oocytes were registered 18 hours after oocyte insemination.
Time Frame: 18 hours after insemination
Population: as for outcome 2
Measure: Number; unit: Percentage of fertilized oocytes
Units Other Than Participants: Number of mature oocytes
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of mature oocytes) | 33 | 23
Percentage of fertilized oocytes | 100 | 33.3
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.480, Chi-squared

8. Secondary Outcome: Number of Cycles With Embryo Transfer (ET)
Description: One or 2 embryos were transferred on day 3 after egg collection. This outcome represents the number of cycles that culminate with embryo transfer.
Time Frame: On day 3 after egg collection
Population: as for outcome 2
Measure: Count of Units; unit: Number of IVF cycles
Units Other Than Participants: Number of IVF cycles
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of IVF cycles) | 16 | 15
Number of IVF cycles | 8 | 4
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.236, Chi-squared

9. Secondary Outcome: Number and Percentage of Cycles With Clinical Pregnancy
Description: Clinical pregnancy was defined as the presence of a gestational sac and heart beat under ultrasonography
Time Frame: 6 weeks after embryo transfer
Population: as for outcome 2
Measure: Count of Units; unit: Number of IVF cycles
Units Other Than Participants: Number of IVF cycles
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Number analyzed (Number of IVF cycles) | 16 | 15
Number of IVF cycles | 3 | 2
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.684, Chi-squared; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.13 to 3.68]

10. Secondary Outcome: Live Birth Rate
Description: Live birth rate was calculated by dividing the number of patients who achieved live birth in each cycle by the number of patients who initiated that cycle
Time Frame: 9 months or birth of one or more live babies
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Experimental Arm
Number analyzed (Participants) | 16 | 15
Participants | 3 | 1
Statistical Analysis 1: Comparison: Control Arm vs Experimental Arm; Test type: Superiority; p = 0.512, Chi-squared; Risk Ratio (RR) = 0.36, 95% CI 2-sided [0.04 to 3.05]

ADVERSE EVENTS:
Time Frame: Day 1 (recruitment) up to final follow-up (6 months after recruitment)
Description: No serious adverse events were registered. Just a postsurgical complication consisting of a 2-day fever episode was registered in 1 patient.
Arm/Group | Control Arm | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=16) | Experimental Arm (N=15)
Minor postsurgical complication (General disorders) | 0 (0) | 1 (1) — After surgery, 1 patient experienced a 2-day episode of fever of unknown origin. She was treated with paracetamol without requiring antibiotic treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT02354963/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT02354963/SAP_001.pdf